CLINICAL TRIAL: NCT02626390
Title: How do Different Styles of Information Provision Affect Learning During Early Gait Training Post Stroke? A Feasibility Study
Brief Title: Information Provision During Early Gait Training Post Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7938
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implicit Learning (Experimental): Physiotherapy delivered based on implicit treatment guidance - achieved primarily by reducing the frequency of verbal coaching statements and promoting an external focus of attention.
  Interventions: Other: Minimal instructions/feedback and an External Focus of Attention
- Explicit Learning (Active Comparator): Physiotherapy delivered based on explicit treatment guidance - achieved primarily by giving frequent verbal coaching statements and promoting an internal focus of attention.
  Interventions: Other: Frequent instructions/feedback and an Internal Focus of Attention

INTERVENTIONS:
Other: Frequent instructions/feedback and an Internal Focus of Attention
  Arms: Explicit Learning
Other: Minimal instructions/feedback and an External Focus of Attention
  Arms: Implicit Learning

SUMMARY:
This study examined the feasibility of using implicit and explicit learning approaches during gait rehabilitation in the early phase following stroke. It was a double blind trial (participants and assessors) using a matched pairs design. Participants were recruited from an acute stroke unit, and were randomised to receive gait rehabilitation over three consecutive days using either an implicit or explicit approach. Guidelines for each were developed empirically, including differences in the amount, timing, and attentional focus of therapists' verbal communication. Sessions were recorded and their content analysed to establish concordance with the guidance. Clinical measures were taken at baseline and 24 hours post intervention using the Berg Balance Scale and the Step Test. Therapists were able to adhere to the guidance. Both approaches were found to be acceptable to both patients and therapists. The findings will be used to design an appropriately powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving rehabilitation for their first episode of stroke which resulted in hemiplegia
* Able to give informed consent to take part in the study.
* Currently receiving physiotherapy for the re-education of gait (at minimum is able to stand, weight bear and take one step with assistance of one person).

Exclusion Criteria:

* Patients with a history of:

  * any other neurological conditions including previous stroke
  * any pre-stroke musculoskeletal condition that either: i. limited walking to less than 100 metres and/or ii. resulted in a noticeable gait abnormality and/or iii. required use of a bilateral walking aid (e.g. 2 walking sticks or a walking frame)
* Patients with marked receptive dysphasia (not able to follow 3-stage commands) - confirmed through liaison with multi-disciplinary team, including Speech and Language Therapists where necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 24 hours post final treatment session

SECONDARY OUTCOMES:
Step Test | 24 hours post final treatment session

IPD SHARING:
Plan to Share IPD: No